CLINICAL TRIAL: NCT04656379
Title: The Incidence and Risk Factors of Postoperative Delirium in Elderly Patients Undergoing Spine Surgery
Brief Title: The Incidence and Risk Factors of Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, PhD, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: delirium_risk factors
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Delirium in Old Age
Keywords: postoperative delirium; elderly; spine surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: spine surgery — Risk factors for postoperative delirium in elderly patients underwent spine surgery will be evaluated.

SUMMARY:
Delirium is known to be one of the most common postoperative complications in elderly patients undergoing surgery. Because postoperative delirium can affect the length of hospital stay and prognosis significantly, it is important to identify the risk factors for postoperative delirium in advance. However, there have been few reports concerning intraoperative modifiable risk factors, such as postoperative pain, for postoperative delirium.

DETAILED DESCRIPTION:
In this observational study, we will review the electronic medical records of elderly patients underwent spine surgery and assess the incidence and risk factors for postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent spine surgery between September 2016 and August 2018 at Seoul National University Hospital

Exclusion Criteria:

* Patients who had no information on postoperative care and managements.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥65 and underwent spine surgery between September 2016 and August 2018 at Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | through study completion, postoperative period up to 2 years after surgery
  Incidence of delirium after spine surgery

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided